CLINICAL TRIAL: NCT01822327
Title: Treating Cocaine Abuse: A Behavioral Approach
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stephen T. Higgins, Professor of Psychiatry and Psychology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA009378 (NIH)
Record Dates: First submitted 2013-02-26; First posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Contingent Vouchers Unmatched (Experimental): CRA therapy plus Voucher incentives contingent on cocaine abstinence with monetary values set at usual monetary values across all patients.
  Interventions: Behavioral: Contingency Management
- Contingent Vouchers, Matched (Experimental): CRA therapy plus Vouchers contingent on cocaine abstinence, with more severe patients receiving twice the usual voucher monetary values.
  Interventions: Behavioral: Contingency Management
- Non-Contingent Vouchers control (Active Comparator): CRA therapy plus Vouchers earned independent of drug use
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — CRA plus Vouchers contingent on drug abstinence with values the same across all patients
  Arms: Contingent Vouchers Unmatched
Behavioral: Contingency Management — CRA plus Vouchers contingent on cocaine abstinence with more severe patients receiving greater value vouchers
  Arms: Contingent Vouchers, Matched
Behavioral: Contingency Management — CRA plus Vouchers earned independent of cocaine use
  Arms: Non-Contingent Vouchers control

SUMMARY:
This study is designed to advance our development of a treatment for cocaine dependence. The investigators hypothesize that clients with high-risk characteristics will benefit from enhanced levels of treatment.

DETAILED DESCRIPTION:
Treatment development for cocaine dependence often proceeds without effort to adapt treatment parameters to patient characteristics. Such a one-size-fits-all approach is problematic because of the heterogeneity of the clinical population. Additionally, the approach is often subject to opposing biases either towards constraining costs or maximizing efficacy. This project includes two sequential clinical trails examining variations of the CRA + Vouchers treatment for cocaine dependence that are designed to explore matching treatment parameters to patient baseline characteristics known to moderate treatment response among cocaine-dependent outpatients. In Trial 1, all patients were randomly assigned to receive 24 weeks of CRA therapy but randomly assigned to one of three voucher-based incentive conditions: (a) 6 weeks of vouchers contingent on abstinence and incentive monetary value at usual level; (b) 6 weeks of vouchers contingent on abstinence but incentive value set at usual level for low-severity patients (intranasal cocaine users or married patients) and at twice the usual value for high severity patients (i.e., unmarried cocaine smokers/injectors), or to (c) a control condition where incentives were provided independent of recent cocaine use. In Trial 2, all patients receive 12 weeks of abstinence-contingent incentives, but randomly assigned to also receive (a) 24 weeks of CRA therapy or (b) 4 weeks of CRA therapy. The overarching goal of the two trials is to strike a balance between the aforementioned biases towards constraining costs or maximizing efficacy and thereby facilitate cost containment without compromising efficacy, especially among more severe patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Meets DSM IV criteria for cocaine dependence

Exclusion Criteria:

* Psychosis
* Pregnancy
* Leaving immediate geographic area sooner than 6 months
* An organic psychiatric disorder
* Medical illness such that participation is not feasible (e.g., on dialysis).
* Subjects in acute alcohol withdrawal
* Uncontrolled seizure disorder
* Significant depression or suicidal ideation (pending psychological evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2007-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Biochemically-Verified Cocaine Use | 2 years

SECONDARY OUTCOMES:
Addiction Severity Inventory Scores | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Higgins, Ph.D, Principal Investigator — University of Vermont
Locations (1):
- Substance Abuse Treatment Center, University of Vermont; UHC, Burlington, Vermont, United States

REFERENCES:
- [Background] Garcia-Rodriguez O, Secades-Villa R, Higgins ST, Fernandez-Hermida JR, Carballo JL. Financing a voucher program for cocaine abusers through community donations in Spain. J Appl Behav Anal. 2008 Winter;41(4):623-8. doi: 10.1901/jaba.2008.41-623. PMID 19192866
- [Background] Higgins, S.T., Heil, S.H., Rogers, R.E., & Chivers, L. (2008). Cocaine. In S.T. Higgins, K. Silverman, & S.H. Heil (Eds.), Contingency management in substance abuse treatment (pp. 19-410. New York, NY: The Guilford Press.
- [Background] Higgins, S.T., Sigmon, S.C., Heil, S.H. (2008). Drug abuse and dependence. In D.H. Barlow (Ed.), Clinical handbook of psychological disorders (4th ed.). (pp. 547-577). New York: Guilford Publications, Inc.
- [Background] Higgins, S.T. & Silverman, K., (2008). Contingency Management. In M. Galanter and H.D. Kleber (Eds.) Textbook of substance abuse treatment (4th ed.). (pp. 387-399). The American Psychiatric Press..
- [Background] Higgins, S.T. & Silverman, K. (2008). Introduction. In S.T. Higgins, K. Silverman, & S.H. Heil (Eds.), Contingency management in substance abuse treatment (pp. 1-15). New York, NY: The Guilford Press.
- [Background] Rogers RE, Higgins ST, Silverman K, Thomas CS, Badger GJ, Bigelow G, Stitzer M. Abstinence-contingent reinforcement and engagement in non-drug-related activities among illicit drug abusers. Psychol Addict Behav. 2008 Dec;22(4):544-50. doi: 10.1037/0893-164X.22.4.544. PMID 19071979
- [Background] Silverman K, Roll JM, Higgins ST. Introduction to the special issue on the behavior analysis and treatment of drug addiction. J Appl Behav Anal. 2008 Winter;41(4):471-80. doi: 10.1901/jaba.2008.41-471. PMID 19192853
- [Background] Garcia-Rodriguez O, Secades-Villa R, Higgins ST, Fernandez-Hermida JR, Carballo JL, Errasti Perez JM, Al-halabi Diaz S. Effects of voucher-based intervention on abstinence and retention in an outpatient treatment for cocaine addiction: a randomized controlled trial. Exp Clin Psychopharmacol. 2009 Jun;17(3):131-8. doi: 10.1037/a0015963. PMID 19586227
- [Background] Higgins ST. Comments on contingency management and conditional cash transfers. Health Econ. 2010 Oct;19(10):1255-8. doi: 10.1002/hec.1543. PMID 19670269
- [Background] Higgins, S. T., Heil, S. H., & Sigmon, S. C. (2010). Voucher-based contingency management in the treatment of substance use disorders. In G. J. Madden (Ed.), APA Handbook of Behavior Analysis. Washington, DC: American Psychological Association.
- [Result] Higgins, S.T. and Rogers, R.E. (2009). Contingency management and community reinforcement approach. In Peter M. Miller (Ed.). Evidence-based addiction treatment (pp. 249-267). Burlington: Academic Press, Elsevier Inc.
- See also: Substance Abuse Treatment Center — http://www.uvm.edu/~uvmsatc/